CLINICAL TRIAL: NCT06457347
Title: Early Versus Ultra Early Surgical Treatment of Ruptured Intracranial Aneurysms: A Randomized Controlled Trial.
Brief Title: Early Versus Ultra Early Surgical Treatment of Ruptured Intracranial Aneurysms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Revaz Dzhindzhikhadze (Other Government)
Responsible Party: Sponsor-Investigator, Revaz Dzhindzhikhadze, Chief of neurosurgical department, Moscow Regional Research and Clinical Institute (MONIKI)
Organization: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sah_moniki
Record Dates: First submitted 2024-05-25; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: aneurysm; subarachnoid hemorrhage; clipping; microsurgery; surgery timing
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra early (<24 hours) (Experimental)
  Interventions: Procedure: Ultra early (<24 hours) ruptured aneurysm clipping
- Early (24-72 hours) (Active Comparator)
  Interventions: Procedure: Early (24-72 hours) ruptured aneurysm clipping

INTERVENTIONS:
Procedure: Ultra early (<24 hours) ruptured aneurysm clipping — Aneurysms are clipped with open surgery in less than 24 hours after rupture to prevent early rebleeding.
  Arms: Ultra early (<24 hours)
Procedure: Early (24-72 hours) ruptured aneurysm clipping — Aneurysms are clipped with open surgery in 24 to 72 hours after rupture to prevent early rebleeding.
  Arms: Early (24-72 hours)

SUMMARY:
The goal of this clinical trial is to determine the most effective timing for clipping in adults with ruptured intracranial aneurysms. It will also assess the safety of performing the surgery at different times of early period after the aneurysm has ruptured. The main questions it aims to answer are:

1. Does ultra-early surgical intervention ( less than 24 hours of rupture) improve survival rates compared to delayed surgery (24 to 72 hours after rupture)?
2. What are the complication rates associated with early versus delayed surgical intervention?

Researchers will compare clipping in ultra-early period to surgery in early period to see if timing affects the outcomes for treating ruptured intracranial aneurysms.

Participants will:

* Be randomly assigned to undergo surgical clipping either within 24 hours of rupture or between 24 hours to 72 hours after the rupture.
* Visit the clinic for follow-up assessments at 1 month, 3 months, 6 months, and 12 months post-surgery.
* Keep a diary of their symptoms, neurological function, and any complications they experience post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* aneurysmal subarachnoid hemorrhage
* patient eligible for surgical clipping
* patients with informed consent for inclusion into the study

Exclusion Criteria:

* patients admitted and treated >72 h after subarachnoid hemorrhage onset
* patients with severe comorbidities
* patients with multiple aneurysms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rebleeding rate before anerysm clipping | baseline, pre-surgery
  The rate of recurrent aneurysm rupture and subarachnoid hemorrhage before aneurysm surgery is performed.

SECONDARY OUTCOMES:
Clinical outcome according to the Modified Rankin Scale | Up to 12 months after aneurysm surgery
  Modified Rankin Scale (mRS) is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0 to 6, spanning from perfect health without symptoms to death:
  0: No symptoms.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead.
Delayed cerebral ischemia | Up to 3 weeks after aneurysm rupture
  Delayed cerebral ischemia is defined as a clinical deterioration attributed to cerebral ischemia that occurs days after an initial subarachnoid hemorrhage. This condition is characterized by a new onset of focal neurological impairment or a decrease of at least two points on the Glasgow Coma Scale, which cannot be attributed to other causes such as rebleeding, hydrocephalus, or surgical complications. The risk of delayed cerebral ischemia is lower when aneurysms are treated in less than 24 h after rupture
Rate of occlusion according to modified Raymond-Roy classification | Up to 12 months after aneurysm surgery
  Modified Raymond-Roy Classification (mRRC) categorizes the occlusion status of an aneurysm post-treatment into three grades based on the extent of filling within the aneurysm sac seen on angiographic imaging:
  Class 1 (Complete Occlusion): No opacification of the aneurysm sac is visible. This indicates a complete absence of blood flow into the aneurysm.
  Class 2 (Residual Neck): A small residual contrast filling is confined to the neck of the aneurysm.
  Class 3 (Residual Aneurysm): There is opacification of the aneurysm sac, indicating incomplete occlusion with more substantial contrast filling.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips TJ, Dowling RJ, Yan B, Laidlaw JD, Mitchell PJ. Does treatment of ruptured intracranial aneurysms within 24 hours improve clinical outcome? Stroke. 2011 Jul;42(7):1936-45. doi: 10.1161/STROKEAHA.110.602888. Epub 2011 Jun 16. PMID 21680909
- [Background] Tan H, Huang G, Li Z, Feng H, Wang Z, Zhao D, Tang J, Liu J. The impact of surgical timing on the management of aneurysms with acute hydrocephalus after aneurysmal subarachnoid hemorrhage. Turk Neurosurg. 2014;24(3):385-90. doi: 10.5137/1019-5149.JTN.9484-13.0. PMID 24848179
- [Background] Oudshoorn SC, Rinkel GJ, Molyneux AJ, Kerr RS, Dorhout Mees SM, Backes D, Algra A, Vergouwen MD. Aneurysm treatment <24 versus 24-72 h after subarachnoid hemorrhage. Neurocrit Care. 2014 Aug;21(1):4-13. doi: 10.1007/s12028-014-9969-8. PMID 24639201
- [Background] Dalbayrak S, Altas M, Arslan R. The effects of timing of aneurysm surgery on vasospasm and mortality in patients with subarachnoid hemorrhage. Acta Neurol Belg. 2011 Dec;111(4):317-20. PMID 22368972
- [Background] Ross N, Hutchinson PJ, Seeley H, Kirkpatrick PJ. Timing of surgery for supratentorial aneurysmal subarachnoid haemorrhage: report of a prospective study. J Neurol Neurosurg Psychiatry. 2002 Apr;72(4):480-4. doi: 10.1136/jnnp.72.4.480. PMID 11909907
- [Background] Dorhout Mees SM, Molyneux AJ, Kerr RS, Algra A, Rinkel GJ. Timing of aneurysm treatment after subarachnoid hemorrhage: relationship with delayed cerebral ischemia and poor outcome. Stroke. 2012 Aug;43(8):2126-9. doi: 10.1161/STROKEAHA.111.639690. Epub 2012 Jun 14. PMID 22700527